CLINICAL TRIAL: NCT04788420
Title: Influence of Co-existing Mutations on Sorafenib Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation for Patients With FLT3-ITD Positive Acute Myeloid Leukemia
Brief Title: Influence of Co-existing Mutations on Sorafenib Maintenance Therapy After Allo-HSCT for Patients With FLT3-ITD AML
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other); Xiangya Hospital of Central South University (Other); First People's Hospital of Chenzhou (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); The First Affiliated Hospital of Soochow University (Other); Xinqiao Hospital of Chongqing (Other); First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: Sorafenib-Flt3 AML-2020
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia With FLT3/ITD Mutation; Hematopoietic Stem Cell Transplantation
Keywords: Acute Myeloid Leukemia; FLT3-ITD; Hematopoietic Stem Cell Transplantation; sorafenib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bone marrow and/or peripheral blood were taken from participants upon enrollment for diagnosis and detection of co-occurring mutations via PCR, direct sequencing and /or new generation sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sorafenib group: Patients assigned to this group received sorafenib post-transplantation.
  Interventions: Drug: Sorafenib
- Control group: Patients assigned to this group did not receive sorafenib or any other FLT3 inhibitor post-transplantation until reaching the primary outcome.

INTERVENTIONS:
Drug: Sorafenib — The initial dose of sorafenib is 400 mg orally twice daily and is adjusted in case of suspected toxicity or resistance (dose range, 200-800 mg daily).
  Other Names: Nexavar; BAY 43-9006; BAY-673472; BAY 545-9085
  Groups: Sorafenib group

SUMMARY:
The purpose of this study is to reveal the influence of co-existing mutations on the efficacy of sorafenib maintenance after allogeneic hematopoietic stem cell transplantation for patients with FLT3-ITD AML.

DETAILED DESCRIPTION:
Internal tandem duplication of FMS-like tyrosine kinase 3 (FLT3-ITD) mutations have been reported in 20%-30% of patients with acute myeloid leukemia (AML). FLT3-ITD-positive AML patients have an inferior survival, primarily due to lower complete remission (CR) rate and higher relapse rate. Our previous studies demonstrated that post-transplantation sorafenib maintenance could improve the outcomes of FLT3-ITD-positive AML patients. However, whether other co-existing mutations influence the efficacy of post-allo-HSCT sorafenib maintenance remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* FLT3-ITD Positive AML
* Allo-HSCT Recipients

Exclusion Criteria:

* cardiac dysfunction (particularly congestive heart failure)
* hepatic abnormalities (bilirubin ≥ 3 mg/dL, aminotransferase> 2 times the upper limit of normal)
* renal dysfunction (creatinine clearance rate < 30 mL/min)
* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (according to the investigators' decision)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cases included in this study were from 4 previously published studies of our study group, including 3 retrospective and 1 prospective studies.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of leukemia relapse | 2 year

SECONDARY OUTCOMES:
Overall survival | 2 year
Leukemia-free survival | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Xuan L, Wang Y, Huang F, Jiang E, Deng L, Wu B, Fan Z, Liang X, Xu N, Ye J, Lin R, Yin C, Zhang Y, Sun J, Han M, Huang X, Liu Q. Effect of sorafenib on the outcomes of patients with FLT3-ITD acute myeloid leukemia undergoing allogeneic hematopoietic stem cell transplantation. Cancer. 2018 May 1;124(9):1954-1963. doi: 10.1002/cncr.31295. Epub 2018 Mar 6. PMID 29509276
- [Background] Xuan L, Wang Y, Huang F, Fan Z, Xu Y, Sun J, Xu N, Deng L, Li X, Liang X, Luo X, Shi P, Liu H, Wang Z, Jiang L, Yu C, Zhou X, Lin R, Chen Y, Tu S, Huang X, Liu Q. Sorafenib maintenance in patients with FLT3-ITD acute myeloid leukaemia undergoing allogeneic haematopoietic stem-cell transplantation: an open-label, multicentre, randomised phase 3 trial. Lancet Oncol. 2020 Sep;21(9):1201-1212. doi: 10.1016/S1470-2045(20)30455-1. Epub 2020 Aug 10. PMID 32791048
- [Background] Xuan L, Wang Y, Chen J, Jiang E, Gao L, Wu B, Deng L, Liang X, Huang F, Fan Z, Tang X, Sun J, Zhang X, Han M, Wu D, Huang X, Liu Q. Sorafenib Therapy Is Associated with Improved Outcomes for FMS-like Tyrosine Kinase 3 Internal Tandem Duplication Acute Myeloid Leukemia Relapsing after Allogeneic Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2019 Aug;25(8):1674-1681. doi: 10.1016/j.bbmt.2019.04.018. Epub 2019 Apr 19. PMID 31009704
- [Background] Shi J, Cao L, Luo Y, Zhao Y, Tan Y, Yu J, Lai X, Zhu Y, Hu Y, He J, Sun J, Zheng W, Wei G, Huang H. Maintenance sorafenib is superior to prophylactic donor lymphocyte infusion at improving the prognosis of acute myeloid leukemia with FMS-like tyrosine kinase 3 internal tandem duplication after allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2021 Jan;56(1):293-296. doi: 10.1038/s41409-020-01015-w. Epub 2020 Aug 4. No abstract available. PMID 32753705